CLINICAL TRIAL: NCT04256499
Title: Water Load Test Value for Hyponatremia Due to a Syndrome of Inappropriate Antidiuresis (SIAD)
Brief Title: Water Load Test Value for Hyponatremia
Acronym: WATERLINE
Status: Completed | Type: Observational
Sponsor: European Georges Pompidou Hospital (Other)
Responsible Party: Principal Investigator, Jean-philippe Bertocchio, MD, PhD, Principal Investigator, European Georges Pompidou Hospital
Other Study IDs: WATERLINE
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: SIAD - Syndrome of Inappropriate Antidiuresis; Hyponatremia
Keywords: hyponatremia; SIAD; water load test
MeSH Terms: conditions — Inappropriate ADH Syndrome; Hyponatremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Water load test: Patients experiencing a syndrome of inappropriate antidiuresis who had an acute water load test
  Interventions: Procedure: Acute water load test
- Control group: Patients who had an acute water load test and who did not experience any water homeostasis anomalies
  Interventions: Procedure: Acute water load test

INTERVENTIONS:
Procedure: Acute water load test — The acute water load test consists in administering orally 20 mL/kg (of body weight) of water (ingested in less than 30 min) and then follow (during 4 to 6 hours) blood and urine parameters.

SUMMARY:
Acute water load test has been using to diagnose renal ability to excrete water for decades. Latest recommendations for the diagnosis of hyponatremia do not recommend performing such a test. The investigators aim at, retrospectively, study the value of acute water load test in patients suffering from a syndrome of inappropriate antidiuresis.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old at the time of the test
* affiliated to a social insurance system
* water load test performed at the Renal and Metabolic Diseases Unit of the European George Pompidou Hospital, AP-HP, Paris, France
* between 01/01/2001 and 12/31/2019

Exclusion Criteria:

* hypernatremia and/or polyuria-polydipsia (diabetes insipidus)
* hyponatremia due to a tea and toast syndrome and/or a beer potomania
* hyponatremia due to a high (or normal) osmolality related to diabetes mellitus, hyperproteinemia and/or intoxication
* chronic kidney disease with an estimated glomerular filtration rate (eGFR) by the MDRD formula <60 mL/min/1.73m2
* hyponatremia related to thiazides
* hyponatremia related to an hypovolemic status
* syndrome of inappropriate antidiuresis related to an endocrine disorder (such as hypothyroidism or adrenal insufficiency)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this retrospective study, the included population is composed only with adult patients experiencing a syndrome of inappropriate antidiuresis (SIAD) who were explored by an acute water load test at the Renal and Metabolic Diseases Unit of the European George Pompidou Hospital, Paris, France.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2001-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Natremia | any time after water load test from hour 2 to hour 6
  Plasma sodium concentration (abnormal if <135mM)

SECONDARY OUTCOMES:
Plasma osmolality | any time after water load test from hour 2 to hour 6
  Plasma osmolality (abnormal if <280mOsm/kgH2O)
Excretion of water load | after water load test from hour 0 to hour 6
  Ratio between the excreted water (in urine) volume and the ingested one
Urine osmolality | any time after water load test from hour 2 to hour 6
  Minimum urine osmolality reached

OTHER OUTCOMES:
Body weight | Value at hour 6 versus initial value (hour 0)
  Variation of body weight during the test

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Bertocchio, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- European Georges Pompidou Hospital, APHP, Paris, France

IPD SHARING:
Plan to Share IPD: No